CLINICAL TRIAL: NCT06527599
Title: Screening in Trauma for Opioid Misuse Prevention - an Adaptive Intervention (STOMP-AI)
Brief Title: Screening in Trauma for Opioid Misuse Prevention - an Adaptive Intervention
Acronym: STOMP-AI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Wisconsin Partnership Program (Other); Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0157; A532050 (Other: UW Madison); Protocol Version CP004 (Other: UW Madison)
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Opioid Misuse; Trauma Injury
MeSH Terms: conditions — Opioid-Related Disorders; Accidental Injuries

STUDY DESIGN:
Intervention Model Description: Pilot Sequential, Multiple-Assignment Randomized Trial (Pilot SMART)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- PCST-Lite + eTCC re-randomized to eTCC + PCST-Plus (Experimental): Participants initially randomized to Pain Coping Skills Training-Lite (PCST-Lite) plus enhanced Trauma Care Coordination (eTCC) who are identified to be at elevated risk for opioid misuse at week 4 may be re-randomized to receive eTCC and Enhanced Pain Coping Skills Training (PCST-Plus).
  Interventions: Other: Opioid Risk Monitoring (ORM); Behavioral: enhanced Trauma Care Coordination (eTCC); Behavioral: Pain Coping Skills Training - Brief (PCST-LITE); Behavioral: Pain Coping Skills Training - Plus (PCST+)
- PCST-Lite + eTCC re-randomized to eTCC + PCST-M (Experimental): Participants initially randomized to PCST-Lite plus eTCC who are identified to be at elevated risk for opioid misuse at week 4 may be re-randomized to receive eTCC and Pain Coping Skills Training-Maintenance (PCST-M) at 4 weeks.
  Interventions: Other: Opioid Risk Monitoring (ORM); Behavioral: enhanced Trauma Care Coordination (eTCC); Behavioral: Pain Coping Skills Training - Brief (PCST-LITE); Behavioral: Pain Coping Skills Training - Maintenance (PCST-M)
- PCST-Lite + eTCC Low Risk eTCC + PCST-M (Experimental): Participants initially randomized to PCST-Lite plus eTCC who are identified to be at low risk for opioid misuse at week 4 will then receive eTCC and PCST-M.
  Interventions: Other: Opioid Risk Monitoring (ORM); Behavioral: enhanced Trauma Care Coordination (eTCC); Behavioral: Pain Coping Skills Training - Brief (PCST-LITE); Behavioral: Pain Coping Skills Training - Maintenance (PCST-M)
- eTCC re-randomized to PCST-LITE (Experimental): Participants initially randomized to eTCC who are identified to be at elevated risk for opioid misuse at week 4 may be re-randomized to PCST-LITE at 4 weeks.
  Interventions: Other: Opioid Risk Monitoring (ORM); Behavioral: enhanced Trauma Care Coordination (eTCC); Behavioral: Pain Coping Skills Training - Brief (PCST-LITE)
- eTCC re-randomized to eTCC (Experimental): Participants initially randomized to eTCC who are identified to be at elevated risk for opioid misuse at week 4 may be re-randomized to receive the same intervention at 4 weeks.
  Interventions: Other: Opioid Risk Monitoring (ORM); Behavioral: enhanced Trauma Care Coordination (eTCC)
- eTCC Low Risk eTCC (Experimental): Participants initially randomized to eTCC who are identified to be at low risk for opioid misuse at week 4 will continue eTCC.
  Interventions: Other: Opioid Risk Monitoring (ORM); Behavioral: enhanced Trauma Care Coordination (eTCC)
- PSCT-LITE re-randomized to PCST+ (Experimental): Participants initially randomized to PCST-LITE who are identified to be at elevated risk for opioid misuse at week 4 re-randomized to PCST+.
  Interventions: Other: Opioid Risk Monitoring (ORM); Behavioral: Pain Coping Skills Training - Brief (PCST-LITE); Behavioral: Pain Coping Skills Training - Plus (PCST+)
- PCST-LITE re-randomized to PCST-Maintenance (Experimental): Participants initially randomized to PCST-LITE and are not re-randomized to an augmented form of PCST will instead receive PCST-Maintenance (PCST-M).
  Interventions: Other: Opioid Risk Monitoring (ORM); Behavioral: Pain Coping Skills Training - Brief (PCST-LITE); Behavioral: Pain Coping Skills Training - Maintenance (PCST-M)
- PCST-Lite Low Risk PCST-M (Experimental): Participants initially randomized to PCST-Lite who are identified to be at low risk for opioid misuse at week 4 will be assigned to PCST-M.
  Interventions: Other: Opioid Risk Monitoring (ORM); Behavioral: Pain Coping Skills Training - Maintenance (PCST-M)
- sTCC re-randomized to PCST-LITE (Experimental): Participants initially randomized to Standard Trauma Care Coordination (sTCC) who are identified to be at elevated risk for opioid misuse at week 4 will be re-randomized to either PCST-LITE or continued sTCC.
  Interventions: Other: Opioid Risk Monitoring (ORM); Behavioral: Pain Coping Skills Training - Brief (PCST-LITE); Behavioral: Standard Trauma Care Coordination (sTCC)
- sTCC re-randomized to sTCC (Experimental): Participants initially randomized to sTCC who are identified to be at elevated risk for opioid misuse at week 4 will be re-randomized to either PCST-LITE or continued sTCC.
  Interventions: Other: Opioid Risk Monitoring (ORM); Behavioral: Standard Trauma Care Coordination (sTCC)
- sTCC Low Risk sTCC (Active Comparator): Participants initially randomized to sTCC who are identified to be at low risk for opioid misuse at week 4 will continued sTCC.
  Interventions: Other: Opioid Risk Monitoring (ORM); Behavioral: Standard Trauma Care Coordination (sTCC)

INTERVENTIONS:
Other: Opioid Risk Monitoring (ORM) — A brief battery of self-reported screeners for risk factors associated with opioid misuse (e.g., Current Opioid Misuse Measure; Pain, Enjoyment of life, and General activities scale; Pain Catastrophizing Scale). These measures will be administered within seven days of hospital discharge (i.e., baseline), and again at 2-, 4-, 8-, and 12-weeks following discharge to assess for ongoing risk for opioid misuse. Participants will additionally complete the self-reported Opioid Risk Tool within seven days of hospital discharge.
Behavioral: enhanced Trauma Care Coordination (eTCC) — An enhanced care management model with increased patient contact and embedded interventions based on clinical presentation and collaboration with the patient. eTCC is a telehealth-based care coordinating intervention where a care coordinator assesses the participant, creates a plan of care, collaborates with the eTCC team, follows up with a second virtual visit within a week, and communicates with the participant and care team at least bi-weekly for the 3 month intervention period.
  Other Names: Trauma Medical Home
  Arms: PCST-Lite + eTCC Low Risk eTCC + PCST-M; PCST-Lite + eTCC re-randomized to eTCC + PCST-M; PCST-Lite + eTCC re-randomized to eTCC + PCST-Plus; eTCC Low Risk eTCC; eTCC re-randomized to PCST-LITE; eTCC re-randomized to eTCC
Behavioral: Pain Coping Skills Training - Brief (PCST-LITE) — PCST-LITE will consist of a single 55-minute videoconference session, in which participants will receive brief psychoeducation grounded in gate control theory, progressive muscle relaxation (PMR), and therapist-guided imagery. Participants will be asked to practice PMR and imagery daily and will receive four weeks of regular (4-5 times per week) text messaging as a reminder.
  Arms: PCST-LITE re-randomized to PCST-Maintenance; PCST-Lite + eTCC Low Risk eTCC + PCST-M; PCST-Lite + eTCC re-randomized to eTCC + PCST-M; PCST-Lite + eTCC re-randomized to eTCC + PCST-Plus; PSCT-LITE re-randomized to PCST+; eTCC re-randomized to PCST-LITE; sTCC re-randomized to PCST-LITE
Behavioral: Standard Trauma Care Coordination (sTCC) — Standard Trauma Care Coordination (sTCC) will functionally serve as a treatment-as-usual arm, as it will involve no study intervention.
  Arms: sTCC Low Risk sTCC; sTCC re-randomized to PCST-LITE; sTCC re-randomized to sTCC
Behavioral: Pain Coping Skills Training - Plus (PCST+) — PCST+ will include two videoconferencing sessions, in addition to the first videoconferencing session they previously received. In session 1, participants will be taught an activity/rest cycle to schedule activities, so they are productive while avoiding increasing pain severity due to taking insufficient breaks. Session 2 centers around cognitive restructuring, involving brief psychoeducation and skills development surrounding how participants might recognize the influence that cognitions can have on pain intensity and coping. Participants will receive 3 weekly, 15-minute calls to review skills and problem-solve.
  Arms: PCST-Lite + eTCC re-randomized to eTCC + PCST-Plus; PSCT-LITE re-randomized to PCST+
Behavioral: Pain Coping Skills Training - Maintenance (PCST-M) — PCST-M consists of five weekly booster calls from the patient's study therapist to reinforce the techniques covered in the initial PCST-Lite session.
  Arms: PCST-LITE re-randomized to PCST-Maintenance; PCST-Lite + eTCC Low Risk eTCC + PCST-M; PCST-Lite + eTCC re-randomized to eTCC + PCST-M; PCST-Lite Low Risk PCST-M

SUMMARY:
The primary objective of the present pilot, sequential, multiple-assignment randomized trial (Pilot SMART) is to determine feasibility and acceptability of delivering (from the perspective of the treatment/intervention staff) and receiving (from the perspective of the patient) an adaptive intervention for reducing rates of opioid misuse and preventing development of opioid use disorder in individuals hospitalized for traumatic injury. A complimentary secondary objective is to ensure the feasibility of conducting a future, multi-site, full-scale SMART.

Approximately 107 participants will be enrolled and can expect to be on study for up to 6 months.

DETAILED DESCRIPTION:
The proposed project would be the first clinical trial to assess the feasibility of implementing a preventative treatment design that specifically targets the needs of individuals receiving opioid prescriptions following surgery for traumatic injury. The project will operationalize a standardized approach to screening, treating, and monitoring risk of opioid misuse following traumatic injury. If funded, the project would provide a personalized approach to post-injury monitoring and management through an adaptive intervention designed to target the needs of the individual, rather than implementing a rigid, one-size-fits-all intervention model to prevent opioid misuse.

Approximately 107 participants will be enrolled into the study (approximately 54 participants at UW and 53 participants at MCW). At or very shortly after (within 1-2 days) discharge, participants will be randomized using a 2x2 factorial design to initially receive any one of the following four interventions:

1. standard Trauma Care Coordination (sTCC)
2. sTCC + an abbreviated Pain Coping Skills Training (PCST-Lite)
3. enhanced Trauma Care Coordination (eTCC)
4. eTCC + PCST-Lite

Components of the adaptive intervention will be iteratively refined at various points before, during, and after the pilot SMART in order to maximize feasibility and acceptability.

Primary Objective: Determine the feasibility of delivering an adaptive intervention for reducing rates of opioid misuse and preventing development of opioid use disorder in individuals hospitalized for traumatic injury.

Secondary Objective: Obtain the preliminary data necessary for a successful NIH R01 Application.

Exploratory Objective 1: Identify associations between the interventions delivered and opioid use/misuse.

Exploratory Objective 2: Identify associations between the interventions delivered and the physical, social, and psychological antecedents of opioid misuse.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak, read, and write fluently in English.
* Admission to site hospital for a traumatic injury at time of screening. A traumatic injury is defined as a physical injury with sudden onset requiring immediate medical attention.
* Injury severity score of 9 or greater.
* Meets at least one of the following descriptions below:

  * Received 40 mg morphine milligram equivalent (MME) within 48 hours of pre-screening; or
  * Discharged with a prescription for an opioid medication.
* Expected to be in control of their own medications at the time of discharge from the controlled environment of hospital or short-term rehabilitation.

Exclusion Criteria:

* Inability to provide written consent for any reason.
* Current self-reported diagnosis of cancer with life expectancy less than 12 months at time of screening.
* Current prescription for opioid use disorder (e.g., suboxone, buprenorphine, methadone, naltrexone), with a current diagnosis of opioid use disorder (OUD) (mild or greater) not in remission.
* History of dementing illnesses and other neurodegenerative diseases such as Alzheimer's disease, Parkinson's disease, or vascular dementia.
* Current significant traumatic brain injury (defined as the presence of any intracranial blood on Computed Tomography scan of the head or best Glasgow Coma Scale Score of less than 13 at the time of screening).
* Current spinal cord injury with persistent neurologic deficit at the time of screening.
* Acute stroke immediately prior to/upon admission, or emergent stroke as a new event during hospitalization.
* Any vision or hearing impairments resulting in an inability to complete study procedures.
* Current pregnancy, as indicated by chart review and self-report.
* Involved in any criminal justice proceedings related to illicit substance use at time of screening.
* Incarcerated or in police custody at time of study enrollment.
* Admitted to the hospital with a burn affecting >10% total body surface area, as indicated by chart review.
* Any medical, physical, cognitive, or psychiatric conditions that would limit the participant's ability to provide informed consent or complete study procedures, as determined by study staff and/or investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percent of Target Sample Size Accrued by Study Completion | up to 18 months
  A feasibility goal is to accrue at least 70 percent of the targeted sample size by study completion.
Number of Participants Enrolled | baseline to 4 weeks, baseline to 12 weeks
  Number of participants who enrolled
Number of Participants Retained | 4 weeks, 12 weeks
  Number of participants who completed the study
Acceptability of intervention | 12 weeks
  Participants will complete a qualitative interview regarding their experiences in the study. Responses may be used to guide future related studies.

SECONDARY OUTCOMES:
Incidence of Adverse Events by Grade | up to 6 months
  A safety objective is to evaluate the frequency and severity of adverse events associated with each arm of the intervention. Reported here is incidence of adverse events by grade.

CONTACTS AND LOCATIONS:
Overall Officials: Randy Brown, MD, PhD, Principal Investigator — UW School of Medicine and Public Health
Locations (2):
- United States (2):
  - UW Health, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No